CLINICAL TRIAL: NCT02980458
Title: Characterisation of Relative Bioavailability of a Generic Deferiprone Formulation in Comparison With a Marketed Reference Product in a Single Dose, 2-period-crossover Design Under Fasting Conditions; Controlled, Open, Randomised, no Blinded Study With Bioequivalence Assessment
Brief Title: Characterisation of Relative Bioavailability With Bioequivalence Assessment of Deferiprone Tablets After Oral Single Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SocraTec R&D GmbH (Other)
Collaborators: SocraMetrics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1221def09ct
Record Dates: First submitted 2016-11-22; First posted 2016-12-02 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-11

CONDITIONS: Bioequivalence
Keywords: Healthy; Bioequivalence; Deferiprone
MeSH Terms: interventions — Deferiprone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deferiprone 500 Lipomed film-coated tablets (Experimental): Oral fasted administration of one film-coated tablet of Deferiprone 500 Lipomed film-coated tablets (Lipomed AG, Switzerland), containing 500 mg deferiprone
  Interventions: Drug: Deferiprone 500Mg Tablet
- Ferriprox® film-coated tablets (Active Comparator): Oral fasted administration of one film-coated tablet of Ferriprox® film-coated tablets (Apotex Europe B.V., Germany), containing 500 mg deferiprone
  Interventions: Drug: Deferiprone 500 MG Oral Tablet [Ferriprox]

INTERVENTIONS:
Drug: Deferiprone 500Mg Tablet
  Arms: Deferiprone 500 Lipomed film-coated tablets
Drug: Deferiprone 500 MG Oral Tablet [Ferriprox]
  Arms: Ferriprox® film-coated tablets

SUMMARY:
The present study will be conducted in order to compare the bioavailability of the generic Test product (Deferiprone 500 Lipomed tablets, Lipomed AG, Switzerland) with a marketed Reference product (Ferriprox® film-coated tablets, Apotex Europe B.V., Germany) both containing 500 mg deferiprone. For this issue the pharmacokinetics will be characterised after single dose administration of each one tablet.

DETAILED DESCRIPTION:
The study will be performed in an open-label, randomised (order of treatments), single dose, 2 period cross-over design with a wash out phase of at least three treatment free days between both administrations. Sample collection will be performed over eight hours after fasted administration. This time is considered adequate for the determination of plasma concentration vs. time profiles long enough for reliable estimation of the extent of absorption, i.e. the AUC derived from measurements is expected to cover at least 80% of the AUC extrapolated to infinity for deferiprone

ELIGIBILITY:
Inclusion Criteria:

1. sex: male
2. ethnic origin: Caucasian
3. age: 18 years or older
4. body-mass index (BMI): >=18.5 kg/m² and <= 30.0 kg/m²
5. good state of health
6. non-smoker or ex-smoker for at least 1 month
7. written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

1. existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
2. existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient
3. existing gastrointestinal diseases or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
4. history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
5. known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations
6. subjects with severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
7. heart rate < 50 bpm
8. laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator
9. laboratory values: CRP > 5 mg/L, ASAT > 20 % ULN, ALAT > 10 % ULN, bilirubin > 20 % ULN and creatinine > 0.1 mg/dL
10. positive anti-HIV-test (if positive to be verified by western blot), HBs-AG-test (if positive to be verified by test for HBc-IgM) or anti-HCV-test
11. history of recurrent episodes of neutropenia or history of agranulocytosis
12. acute or chronic diseases which may interfere with the pharmacokinetics of the IMP
13. history of or current drug or alcohol dependence
14. regular intake of alcoholic food or beverages of ≥ 40 g pure ethanol for male per day
15. subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
16. regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
17. blood donation or other blood loss of more than 400 ml within the last 2 months prior to individual enrolment of the subject
18. administration of any investigational medicinal product during the last 2 months prior to individual enrolment of the subject
19. regular treatment with any systemically available medication
20. treatment with medicinal products which might cause neutropenia or agranulocytosis
21. subjects, who report a frequent occurrence of migraine attacks
22. subjects suspected or known not to follow instructions
23. subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC0-tlast) for deferiprone | 8 hours interval
Peak Plasma Concentration (Cmax) for deferiprone | 8 hours interval

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | from fist dose until discharge of the subject (approx. 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius Koch, MD, Principal Investigator — SocraTec R&D GmbH, Clinical Pharmacology Unit
Locations (1):
- SocraTec R&D GmbH Clinical Pharmacology Unit, Erfurt, Thuringia, Germany